CLINICAL TRIAL: NCT03449368
Title: The Impact of Achondroplasia on Quality of Life, Healthcare Resource Use, Clinical, Socio-economic and Psychosocial State of the Individual.
Brief Title: Lifetime Impact of Achondroplasia Study in Europe-LIAISE
Acronym: LIAISE
Status: Completed | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 111-501
Record Dates: First submitted 2017-12-14; First posted 2018-02-28 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2020-02

CONDITIONS: Achondroplasia
MeSH Terms: conditions — Achondroplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Cohort 1: Includes age group 5-10 with a cap at 50 subjects. This is a retrospective, observational study.
- Cohort 2: Includes age group 11-15 with a cap of 50 subjects. This is a retrospective, observational study.
- Cohort 3: Includes age group 16-20 with a cap of 40 subjects. This is a retrospective, observational study.
- Cohort 4: Includes age group 21-30 with a cap of 40 subjects. This is a retrospective, observational study.
- Cohort 5: Includes age group 31-40 with a cap at 40 subjects. This is a retrospective, observational study.
- Cohort 6: Includes age group 41-50 with a cap at 40 subjects. This is a retrospective, observational study.
- Cohort 7: Includes age group 51-70 with a cap at 40 subjects. This is a retrospective, observational study.

SUMMARY:
Observational study looking at the burden of illness in achondroplasia subjects aged 5-70. The study will include a 5 year review of historical clinical data as well as a single point collection of questionnaire data to look at the impact on the following in individuals with achondroplasia versus a normative population:

* Quality of life
* Clinical burden
* Healthcare resource use
* Socio-economic burden
* Psychosocial burden

Up to 300 subjects will be included in sites in Germany, Spain, Italy, Sweden, Austria and Denmark

DETAILED DESCRIPTION:
This is a multinational, epidemiological, observational, retrospective, cross-sectional study of individuals with achondroplasia (subjects). This study will be conducted at up to approximately 20 sites in European countries.

Subjects will be invited to enroll via 3 routes:

1. During routine hospital visits
2. From subject lists of those previously treated but no longer followed at the study site.
3. Through collaboration of the Investigator with achondroplasia patient organizations, other achondroplasia-related organizations, other healthcare professionals in their country and achondroplasia-related social media sites. A recruitment flyer will be provided to these organizations, healthcare professionals and social media sites and will to be distributed to potential subjects.

Data will be collected over a minimum of the five years prior to the date of enrolment. Clinical and healthcare resource use data will be collected from medical records. For each subject enrolled, data from medical records will be collected and entered onto an electronic case report form (eCRF) at each site. Data collection from medical records will be supplemented by records provided by the subject and, if necessary, confirmed by the family doctor.

Data about QoL, psychosocial burden, socioeconomic burden and healthcare resource use will be collected via a booklet of validated and structured questionnaires.

Characteristics of subjects with achondroplasia (QoL scores, healthcare resource use, educational level, family status, employment status) will be compared with those of the general population, where available.

As this is an observational study, participation will not affect the subject/Investigator relationship, nor influence Investigator's treatment, therapeutic or other management of the subject.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with a documented diagnosis of achondroplasia based on:

   1. Genetic confirmation of achondroplasia and/or
   2. Clinical diagnosis of achondroplasia (clinical examination or radiological assessment)
2. ≥ five years of age at the time of enrolment
3. Has the cognitive and linguistic capacities necessary to complete questionnaires in the language of his/her country (and/or parents/legally acceptable representatives, as applicable)
4. Agrees to participate in the study and has read, understood, completed and signed:

   1. Informed Consent Form (ICF) - for adult subjects
   2. Informed Assent Form (IAF) - for minor subjects, accompanied by a parental ICF completed by their parents/legally acceptable representatives. The age at which the minor subjects sign the IAF will be subject to local requirements.
5. Has medical records available for at least the five years prior to the date of enrolment.

Exclusion Criteria:

1. Currently participating, or participated within the last six months, in

   1. a clinical trial of a medicinal product or medical device or,
   2. other non-clinical, low interventional studies
2. Currently participating or participated in any BioMarin study at any time.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a diagnosis of Achondroplasia aged 5 years or older in Sweden, Germany, Spain, Italy, Austria and Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2017-12-17 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Healthcare resource use | Once at start of study per subject through completion of questionnaires and via retrospective review of historical data. These will be assessed at interim analysis November 2018 and again at end of study with final Clinical Study Report March 2020
  Healthcare resource use will be collected from medical records and through patient questionnaires. Data collection from medical records will be supplemented by records provided by the subject and, if necessary, confirmed by the family doctor. Healthcare resource use will be collected via a booklet of validated and structured questionnaires

SECONDARY OUTCOMES:
Socio-economic burden (educational, personal, employment and financial impact) | Outcomes will be collected once at start of study per subject through completion of questionnaires. These will be assessed at interim analysis November 2018 and again at end of study with final Clinical Study Report March 2020
  Data about socio-economic burden will be collected via a booklet of validated and structured questionnaires specifically the Work and Productivity and Activity Impairment (WPAI-SHP)
Pediatric Functional Independence Measure (WeeFIM) | Data will be collected once at start of study per subject through completion of questionnaires. These will be assessed at interim analysis November 2018 and again at end of study with final Clinical Study Report March 2020
  The WeeFIM measures the need for assistance and the severity of disability in children between six months and seven years of age. The instrument consists of 18 items covering three domains: self-care, mobility, and cognition. The mean total score within each domain and the overall total score will be summarized.
Adolescent Pediatric Pain Tool (APPT) | Data will be collected once at start of study per subject through completion of questionnaires. These will be assessed at interim analysis November 2018 and again at end of study with final Clinical Study Report March 2020
  The APPT is an instrument for self-reporting of pain by children and adolescents aged 8-17 years. Five subscale scores will be summarized on the analysis population
Pediatric Quality of Life Inventory (PedsQL) | Data will be collected once at start of study per subject through completion of questionnaires. These will be assessed at interim analysis November 2018 and again at end of study with final Clinical Study Report March 2020
  The PedsQL is comprised of four dimensions: Physical, Emotional, Social, and School Functioning. The overall score for each dimension is defined as the mean score for each item involved in the dimension. The overall score for each dimension and the mean total score across dimensions will be summarized for each report.
Quality of Life Short Stature Youth (QoLiSSY) Questionnaire | Data will be collected once at start of study per subject through completion of questionnaires. These will be assessed at interim analysis November 2018 and again at end of study with final Clinical Study Report March 2020
  The QoLISSY Questionnaire for children and adolescents consists of the core QOL dimensions: Physical, Social and Emotional, and three predictors of quality of life: Coping, Beliefs and Treatment. The QoLISSY total score is calculated by the sum of the means in the physical, social and emotional sub-scales divided by 3.
Nottingham Health Profile(NHP) Questionnaire | Data will be collected once at start of study per subject through completion of questionnaires. These will be assessed at interim analysis November 2018 and again at end of study with final Clinical Study Report March 2020
  The NHP is a generic quality of life survey used to measure subjective physical, emotional, and social aspects of health. The NHP total score is calculated by averaging the six domain scores.
Brief Pain Inventory-Short Form (BPI-SF) Questionnaire | Data will be collected once at start of study per subject through completion of questionnaires. These will be assessed at interim analysis November 2018 and again at end of study with final Clinical Study Report March 2020
  The BPI-SF is used to assess clinical pain. A mean severity score and mean interference score will be calculated and summarized for the analysis population
EuroQol - 5 Dimensions - 5 Levels (EQ-5D-5L) Questionnaire | Data will be collected once at start of study per subject through completion of questionnaires. These will be assessed at interim analysis November 2018 and again at end of study with final Clinical Study Report March 2020
  EQ-5D-5L questionnaire has 5 dimensions: "Mobility", "Human Autonomy," "Current Activities", "Pain / Discomfort", "Anxiety / Depression" and all dimensions are described by 5 problem levels corresponding to patient response choices. A quality of life score is obtained according to the answers to the questionnaires.

OTHER OUTCOMES:
Measurement of Height | Retrospective data will be collected for 5 years prior to date of enrolment
  Height measurements will be collected from retrospective data where available for standing and sitting height measurements. The height data will be measured in centimetres.
Measurement of Weight Body Mass Index | Retrospective data will be collected for 5 years prior to date of enrolment
  Weight will be collected from retrospective data collected and will be entered in kilograms.
Body Mass Index (BMI) | Retrospective data will be collected for 5 years prior to date of enrolment
  Body Mass Index is calculated using height and weight. Body Mass Index (BMI) will be measured in kg/m2

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — BioMarin Pharmaceutical
Locations (13):
- Medizinische Universitat Wien, Vienna, Austria
- Aarhus Universitetshospital, Aarhus, Denmark
- Germany (3):
  - Klinik für Kinder- und Jugendmedizin, Cologne
  - Medizinische Fakultät, Universitätskinderklinik (KPAE), Magdeburg
  - Universitätsmedizin, Mainz
- Italy (3):
  - UOC Pediatria, Como
  - Maternal and Child Health - University of Genova, Genova
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Spain (4):
  - Hospital Universitario La Paz, Madrid
  - Se ubica en los siguientes centros, Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Unidad de Dismorfología y metabolismo Hospital Universitario Virgen del Rocío, Seville
- Karolinska Hospital, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: August 2020

REFERENCES:
- [Derived] Maghnie M, Semler O, Guillen-Navarro E, Selicorni A, Heath KE, Haeusler G, Hagenas L, Merker A, Leiva-Gea A, Gonzalez VL, Raimann A, Rehberg M, Santos-Simarro F, Ertl DA, Gregersen PA, Onesimo R, Landfeldt E, Jarrett J, Quinn J, Rowell R, Pimenta J, Cohen S, Butt T, Shediac R, Mukherjee S, Mohnike K. Lifetime impact of achondroplasia study in Europe (LIAISE): findings from a multinational observational study. Orphanet J Rare Dis. 2023 Mar 15;18(1):56. doi: 10.1186/s13023-023-02652-2. PMID 36922864